CLINICAL TRIAL: NCT05139355
Title: Health Effects of Oat and Oat Bioactive in Human
Brief Title: Health Effects of Oat and Oat Polar Lipids in Human
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Swedish Foundation for Strategic Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: Dnr. 2018/658
Record Dates: First submitted 2021-11-17; First posted 2021-12-01 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Postprandial Glucose Regulation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Oat product 1 (Experimental): The test portion is based on 50 gram available carbohydrates with added vegetable oil A. Test portion consumed as a breakfast meal prior to determinations of test variables in the morning.
  Interventions: Combination Product: Effects of Oat and Oat Components on Cardiometabolic risk variables
- Oat product 2 (Experimental): The test portion is based on 50 gram available carbohydrates with added vegetable oil B. Test portion consumed as a breakfast meal prior to determinations of test variables in the morning.
  Interventions: Combination Product: Effects of Oat and Oat Components on Cardiometabolic risk variables
- Oat product 3 (Experimental): The test portion is based on 50 gram available carbohydrates with added vegetable oil C. Test portion consumed as a breakfast meal prior to determinations of test variables in the morning.
  Interventions: Combination Product: Effects of Oat and Oat Components on Cardiometabolic risk variables
- Control Product (Placebo Comparator): The test portion is based on 50 gram available carbohydrates without added vegetable oil.
  Interventions: Combination Product: Effects of Oat and Oat Components on Cardiometabolic risk variables

INTERVENTIONS:
Combination Product: Effects of Oat and Oat Components on Cardiometabolic risk variables — Oat and oat bioactive components consumed as breakfast meal.

SUMMARY:
Aim of the study is to investigate health effects of oats and oat derived components, in human intervention studies, with the purpose to build new knowledge for development of cardiometabolic protective foods.

DETAILED DESCRIPTION:
The overall goal is to increase the knowledge which can be used for the development of food products with anti-diabetic properties, with the purpose to facilitate healthier food choices for people. More specifically the primary purpose of this project is to evaluate effects in healthy humans on cardiometabolic test markers of oat and oat based product. The new knowledge will form a base for the development of oat based food products with added health values.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adults
* BMI 18.5 - 28 Kg/m2
* Non smokers
* Consuming a non-vegetarian diet that follows the Nordic diet recommendation.

Exclusion Criteria:

* Fasting blood glucose concentration >6.1 mmol/l
* Known cardio-metabolic disease (e.g. diabetes, hypertension, metabolic syndrome).
* Gastro-intestinal disorders such as IBS (irritable bowel syndrome) that can interfere with the study results, food allergies.
* No antibiotics or probiotics should have been consumed within 4 weeks prior to and during the study.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-11-16 (Actual); Primary Completion 2022-02-26 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Blood glucose regulation | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Postprandial blood glucose regulation (incremental area under the curve) acute after intake of the test products and at forthcoming meals within 5.5 hours after consumption of test products.

SECONDARY OUTCOMES:
Serum insulin | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Acute effects of postprandial serum insulin concentrations (incremental area under the curve) after intake of the test products.
plasma GLP-1 (glucagon-like peptide-1 ) | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Gastro-intestinale hormones involved in appetite and metabolic regulation
Serum triglycerides | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Cardiometabolic risk markers
Serum Free Fatty Acids | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Cardiometabolic risk markers
Plasma PYY (peptide tyrosine tyrosine) | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Gastro-intestinale hormones involved in appetite and metabolic regulation

OTHER OUTCOMES:
Subjective appetite sensations | 0 - 5.5 hours ( at fasting and then repeatedly after breakfast and Standardize lunch)
  Determined with VAS (visual analogue scale) scales (0-100 mm) as a range of subjective sensations related to appetite (such as hunger, desire to eat or fullness)

CONTACTS AND LOCATIONS:
Overall Officials: Anne Nilsson, PhD, Principal Investigator — Department of Food Technology, Engineering and Nutrition, Lund Univesity
Locations (1):
- Food Technology, engineering and Nutrition, LTH, Lund University, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hossain MM, Tovar J, Cloetens L, de Kam S, Nilsson A. Oat polar lipids and sunflower lecithin similarly improve cardiometabolic risk markers and appetite controlling hormone responses after breakfast and a subsequent lunch. A randomized crossover study in healthy adults. Front Nutr. 2024 Nov 6;11:1497844. doi: 10.3389/fnut.2024.1497844. eCollection 2024. PMID 39568724